CLINICAL TRIAL: NCT06151171
Title: Pharmacokinetics of Different CoQ10 Formulations - a Randomized, Double-blind, Single-dose, Crossover Study on the Bioavailability
Brief Title: Pharmacokinetics of Different CoQ10 Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Collaborators: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-02-005
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Coenzyme Q10 Pharmacokinetics
Keywords: bioavailability; CoQ10; Ubiquinol; delivery system; pharmacokinetics
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lipomicel Q10 (Experimental): Lipomicel Q10 (Natural Factors, Burnaby, BC, Canada). One soft gel capsule contains: 100 mg ubiquinone (oxidized form of CoQ10)
  Interventions: Dietary Supplement: CoQ10
- CoQ10 NOW® Ubiquinol (Active Comparator): CoQ10 (NOW® Ubiquinol, Bloomingdale, IL, USA). One soft gel capsule contains: 100 mg ubiquinol (reduced form of CoQ10).
  Interventions: Dietary Supplement: CoQ10
- Qunol Ultra CoQ10 (Active Comparator): Qunol Ultra CoQ10 (Quten Research Institute, LLC, USA). One soft gel contains: 100 mg ubiquinone.
  Interventions: Dietary Supplement: CoQ10

INTERVENTIONS:
Dietary Supplement: CoQ10 — Participants will be randomly and blindly assigned to receive a single dose (200 mg) of one of the preparations (treatments).
  Fasting blood samples are taken at baseline (t=0) or pre-dose for CoQ10 baseline determination.
  Participants receive treatment at time zero with a glass of water (~ 125 mL), along with a standardized breakfast-provided immediately after the dose.
  Capsules are administered as a single oral dose, with a wash-out period of at least 3-4 weeks between the two Coenzyme Q10 test products.
  Capillary blood samples are collected at time points 0, 0.5, 1, 2, 3, 4,5, 6, 8, 10, 12, 24, 48- and 72-hours post-dose. A standardized lunch is provided after the 4hr blood sample, as well as a standardized dinner after the 8-h sample. Identical meals are served to all participants on each test day.

SUMMARY:
The objective of this trial is to compare the bioavailability (AUC, Tmax, and Cmax) of different Coenzyme Q10 preparations in healthy adults. Pharmacokinetic parameters of orally ingested CoQ10 such as AUC, Cmax and Tmax, as well as the ratio of reduced CoQ10 levels to total CoQ10 plasma levels (using the AUC) after administration are compared.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to meet the following criteria to be eligible for enrollment: male or female aged 21-65 years or older
* Participants must complete an online health questionnaire on their medical history (pregnancy must be excluded) upon study enrolment.
* Voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Unstable medical condition; use of any acute medications during study period.
* Use of Coumadin Warfarin; use of supplements containing Coenzyme Q10, including the intake of any other supplements within 2 weeks of the beginning of the study (except for vitamin D and calcium). The use of any supplements except for vitamin D and calcium, are prohibited for the duration of the study.
* History of serious acute or chronic diseases such as gastrointestinal disorders, liver-, kidney-, cardiovascular, or hematological disease or diabetes; or other diseases; intolerances or food allergies such as gluten (in terms of the standardized meals).
* Using any form of nicotine or tobacco; participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
AUC: (the area under the concentration-time curve) to evaluate the absorption of orally ingested CoQ10 in different formulations and determine the ratio of reduced CoQ10 levels to total CoQ10 concentrations in healthy adults. | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  Blood concentrations of reduced and total CoQ10 are analyzed by ultra-performance liquid chromatography (UHPLC) coupled to a Thermo QExactive Orbitrap Mass Spectrometer.
Cmax: (maximum plasma concentration) To evaluate the peak concentrations of orally ingested CoQ10 in different formulations and determine the ratio of reduced CoQ10 levels to total CoQ10 concentrations in healthy adults. | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
Tmax: (the time point of maximum plasma concentration) of orally ingested CoQ10 in different formulations and determine the ratio of reduced CoQ10 levels to total CoQ10 concentrations in healthy adults. | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- ISURA, Burnaby, British Columbia, Canada